CLINICAL TRIAL: NCT04752202
Title: The Influence of Reducing Diets on Changes in Thyroid Parameters in Women Suffering From Obesity and Hashimoto's Disease
Brief Title: The Influence of Reducing Diets on Changes in Thyroid Parameters in Obese Women With Hashimoto's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R-I-002/187/2019
Record Dates: First submitted 2021-02-02; First posted 2021-02-12 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Hashimoto Disease; Obesity
Keywords: Hashimoto; Obesity; Elimination diet; Thyroid gland; Adults
MeSH Terms: conditions — Hashimoto Disease; Obesity; Thyroid Diseases | interventions — Diet, Reducing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (group A) (Experimental): The women were randomly assigned to group A. Test group included 50 women aged 18-65 years with previously diagnosed Hashimoto's disease and obesity. Hashimoto's disease (AITD) was diagnosed by a specialist based on the ultrasound image characteristic of AITD and high levels of anti-thyroid antibodies.
  Interventions: Behavioral: Individually balanced elimination/reducing diets
- Control group (group B) (Other): The women were randomly assigned to group B. Control group included 50 women aged 18-65 years with previously diagnosed Hashimoto's disease and obesity. Hashimoto's disease (AITD) was diagnosed by a specialist based on the ultrasound image characteristic of AITD and high levels of anti-thyroid antibodies.
  Interventions: Behavioral: Individually balanced reducing diets (without elimination)

INTERVENTIONS:
Behavioral: Individually balanced elimination/reducing diets — Participants received diets in the range of 1400-1600 kcal/day (with a deficit of about 1000 kcal/day, depending on the resting metabolism and energy expenditure during the day). At the initial visit and every subsequent month, the women received individually balanced elimination/reducing diets, in accordance with the previously performed food sensitivity tests for 6 months. Laboratory tests for type III food sensitivity in the IgG1-3 class using the ELISA method were performed in an accredited medical laboratory. Diets were designed by a qualified dietitian using the Aliant (Poland) diet calculator. Each diet had the same macronutrient content - 25% protein, 30% fat, and 45% carbohydrate, and met the daily requirements for micro and macro elements for the given age group.
  Arms: Test group (group A)
Behavioral: Individually balanced reducing diets (without elimination) — Participants received diets in the range of 1400-1600 kcal/day (with a deficit of about 1000 kcal/day, depending on the resting metabolism and energy expenditure during the day). At the initial visit and every subsequent month, the women received individually balanced reducing diets (without elimination) for 6 months.Diets were designed by a qualified dietitian using the Aliant (Poland) diet calculator. Each diet had the same macronutrient content - 25% protein, 30% fat, and 45% carbohydrate, and met the daily requirements for micro and macro elements for the given age group.
  Arms: Control group (group B)

SUMMARY:
Hashimoto's disease is listed among the most common endocrine causes of obesity. As treatment of obesity in women with Hashimoto's disease is frequently unsuccessful, the aim of this study was to evaluate the effectiveness of two different reducing diets and their influence on changes in thyroid parameters in the female patients. A six-month observational/interventional study was performed on 100 women aged 18-65 years, previously diagnosed with Hashimoto's disease and obesity and receiving L-thyroxine. The women were randomly assigned to the test group (group A, n=50) following elimination/reducing diets, and the control group (group B, n=50) following reducing diets with the same caloric content (without elimination). Anthropometric and thyroid parameters were evaluated at the beginning, after 3 months and after 6 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Hashimoto's disease
* BMI over 30 kg/m2
* Taking the L-thyroxine, 200 mcg of 1-selenomethionine/day, and 30 mg of zinc gluconate/day throughout the study period

Exclusion Criteria:

---

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Effect of reducing/elimination diets based on IgG1-3 food sensitivity tests and standard balanced reducing diets on body weight changes in patients from obesity and Hashimoto's disease. | This measurement was repeated during 3 visits every 12 weeks.
  The body weight (kg) was measured using a scale with a stadiometer.
Effect of reducing/elimination diets based on IgG1-3 food sensitivity tests and standard balanced reducing diets on body weight changes in patients suffering from obesity and Hashimoto's disease. | This measurement was repeated during 3 visits every 12 weeks.
  The height (cm) was measured using a scale with a stadiometer. This measurement is needed to calculate the Body Mass Index.
Effect of reducing/elimination diets based on IgG1-3 food sensitivity tests and standard balanced reducing diets on Body Mass Index changes in patients suffering from obesity and Hashimoto's disease. | This measurement was repeated during 3 visits every 12 weeks.
  Body Mass Index (kg/m^2) was calculated from the measurements of height and weight using a mathematical formula.
Effect of reducing/elimination diets based on IgG1-3 food sensitivity tests and standard balanced reducing diets on changes in muscle mass in patients suffering from obesity and Hashimoto's disease. | This measurement was repeated during 3 visits every 12 weeks.
  Muscle mass (kg) was determined using the bioimpedance method with a TANITA BC-420 body composition analyzer (T6360, Japan).
Effect of reducing/elimination diets based on IgG1-3 food sensitivity tests and standard balanced reducing diets on changes in total body water in patients suffering from obesity and Hashimoto's disease. | This measurement was repeated during 3 visits every 12 weeks.
  Total body water (kg) was determined using the bioimpedance method with a TANITA BC-420 body composition analyzer (T6360, Japan).
Effect of reducing/elimination diets based on IgG1-3 food sensitivity tests and standard balanced reducing diets on changes in percent body fat in patients suffering from obesity and Hashimoto's disease. | This measurement was repeated during 3 visits every 12 weeks.
  Percent body fat (%) was determined using the bioimpedance method with a TANITA BC-420 body composition analyzer (T6360, Japan).
Effect of reducing/elimination diets based on IgG1-3 food sensitivity tests and standard balanced reducing diets on changes in thyroid parameters in patients suffering from obesity and Hashimoto's disease. | This examination was repeated during 3 visits every 12 weeks.
  Laboratory tests were performed to determine the following serum levels: TSH, fT3, fT4, anti-TPO, and anti-TG. Blood samples were collected in an accredited medical laboratory, in the morning, on an empty stomach after a 12-hour fast.
Effect of reducing/elimination diets based on IgG1-3 food sensitivity tests and standard balanced reducing diets on changes in glucose blood level in patients suffering from obesity and Hashimoto's disease. | This examination was repeated during 3 visits every 12 weeks.
  Laboratory tests were performed to determine glucose blood level. Blood samples were collected in an accredited medical laboratory, in the morning, on an empty stomach after a 12-hour fast.
Effect of reducing/elimination diets based on IgG1-3 food sensitivity tests and standard balanced reducing diets on changes in lipid profile in patients suffering from obesity and Hashimoto's disease. | This examination was repeated during 3 visits every 12 weeks.
  Laboratory tests were performed to determine the lipid profile: total cholesterol, high-density lipoprotein (HDL), low-density (LDL) cholesterol and triglycerides. Blood samples were collected in an accredited medical laboratory, in the morning, on an empty stomach after a 12-hour fast.

CONTACTS AND LOCATIONS:
Overall Officials: Lucyna Ostrowska, Professor, Study Director — Medical University of Bialystok; Dominika Gier, PhD, Principal Investigator — Medical University of Bialystok
Locations (1):
- Department of Dietetic and Clinical Nutrition; Medical University of Bialystok, Bialystok, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Song RH, Wang B, Yao QM, Li Q, Jia X, Zhang JA. The Impact of Obesity on Thyroid Autoimmunity and Dysfunction: A Systematic Review and Meta-Analysis. Front Immunol. 2019 Oct 1;10:2349. doi: 10.3389/fimmu.2019.02349. eCollection 2019. PMID 31681268
- [Background] Rotondi M, Leporati P, Rizza MI, Clerici A, Groppelli G, Pallavicini C, La Manna A, Fonte R, Magri F, Biondi B, Chiovato L. Raised serum TSH in morbid-obese and non-obese patients: effect on the circulating lipid profile. Endocrine. 2014 Feb;45(1):92-7. doi: 10.1007/s12020-013-9928-8. Epub 2013 Mar 23. PMID 23526236
- [Background] Moulin de Moraes CM, Mancini MC, de Melo ME, Figueiredo DA, Villares SM, Rascovski A, Zilberstein B, Halpern A. Prevalence of subclinical hypothyroidism in a morbidly obese population and improvement after weight loss induced by Roux-en-Y gastric bypass. Obes Surg. 2005 Oct;15(9):1287-91. doi: 10.1381/096089205774512537. PMID 16259889
- [Background] Draman MS, Stechman M, Scott-Coombes D, Dayan CM, Rees DA, Ludgate M, Zhang L. The Role of Thyrotropin Receptor Activation in Adipogenesis and Modulation of Fat Phenotype. Front Endocrinol (Lausanne). 2017 Apr 19;8:83. doi: 10.3389/fendo.2017.00083. eCollection 2017. PMID 28469599
- [Background] Krysiak R, Okopien B. The effect of levothyroxine and selenomethionine on lymphocyte and monocyte cytokine release in women with Hashimoto's thyroiditis. J Clin Endocrinol Metab. 2011 Jul;96(7):2206-15. doi: 10.1210/jc.2010-2986. Epub 2011 Apr 20. PMID 21508145
- [Background] Carroccio A, D'Alcamo A, Cavataio F, Soresi M, Seidita A, Sciume C, Geraci G, Iacono G, Mansueto P. High Proportions of People With Nonceliac Wheat Sensitivity Have Autoimmune Disease or Antinuclear Antibodies. Gastroenterology. 2015 Sep;149(3):596-603.e1. doi: 10.1053/j.gastro.2015.05.040. Epub 2015 May 27. PMID 26026392
- [Background] Krysiak R, Szkrobka W, Okopien B. The Effect of Gluten-Free Diet on Thyroid Autoimmunity in Drug-Naive Women with Hashimoto's Thyroiditis: A Pilot Study. Exp Clin Endocrinol Diabetes. 2019 Jul;127(7):417-422. doi: 10.1055/a-0653-7108. Epub 2018 Jul 30. PMID 30060266
- [Background] Pandit AA, Vijay Warde M, Menon PS. Correlation of number of intrathyroid lymphocytes with antimicrosomal antibody titer in Hashimoto's thyroiditis. Diagn Cytopathol. 2003 Feb;28(2):63-5. doi: 10.1002/dc.10235. PMID 12561021